CLINICAL TRIAL: NCT02974465
Title: Electromyographic Biofeedback and Physical Therapy in Upper Limb Hemiparesis: A Randomized Controlled Clinical Trial
Brief Title: Electromyographic Biofeedback and Physical Therapy in Upper Limb Hemiparesis
Acronym: EMG-BFB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Cristina Lirio Romero, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIALCALA
Record Dates: First submitted 2016-11-20; First posted 2016-11-28 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2016-11

CONDITIONS: Electromyography
Keywords: Brain injuries; upper extremity; biofeedback; electromyography; recovery of function
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): protocol of Biofeedback Electromyography plus conventional physical therapy treatment
  Interventions: Procedure: Biofeedback Electromyography; Procedure: Conventional Physical Therapy Treatment
- Control Group (Sham Comparator): consisted of Sham- Biofeedback Electromyography plus conventional physical therapy treatment
  Interventions: Procedure: Sham Biofeedback Electromyography; Procedure: Conventional Physical Therapy Treatment

INTERVENTIONS:
Procedure: Biofeedback Electromyography — protocol of sEMG-BFB that consisted of active movements in glenohumeral abduction guided by the visual signal of the register equipment. The protocol was the following: firstly proof active movements were requested in glenohumeral abduction without feeling any pain in order to teach the visual signal of their muscle activity. The therapist dedicated around 10 minutes in each session for subject learned to control the activation of both muscles in the limits that physical therapist marked with each individual in particular (controlling the activation in the upper trapezius). Once integrated information, shoulder abduction were requested following 4 main principles.
  Arms: Experimental Group
Procedure: Sham Biofeedback Electromyography — consisted of Sham-EMG biofeedback, in which the electrodes were placed as the same method as the EG (Fig. 2) but the screen emit no signal. The subject performed 3 sequences of 10 abduction contractions (first degrees) without pain feeling and with 5 minutes of rest between sequences.
  Arms: Control Group
Procedure: Conventional Physical Therapy Treatment — All participants received a conventional daily treatment of neurological physical therapy. Since no evidence has been found about a specific therapy that specially could benefit hemiparesis consequences, the common approach in this center consists of a combination of different specific concepts (Bobath, Brunnstrom, Rood, Johnstone, Propioceptive Neuromuscular Facilitation, Perfetti, Vojta, Motor Relearning Programme,…), exercise programs, electrotherapy, myofascial techniques, etc…

SUMMARY:
The aim of this study was to assess the effect of a specific protocol of sEMG-BFB in upper limb hemiparesis added to conventional physical therapy on changes in upper extremity functionality, motor recruitment pattern and range of motion (ROM) compared to the single application of conventional physical therapy. It aims to find a 22.22% difference between both interventions.

DETAILED DESCRIPTION:
Upper limb hemiparesis is a common consequence after brain damage.

Objective: To evaluate the effect of a specific protocol of surface electromyographic biofeedback (sEMG-BFB) and conventional physical therapy in upper limb functionality, muscle recruitment changes, and glenohumeral range of motion compared to the single application of conventional physical therapy.

Design: randomized controlled clinical trial.

Sample: 40 participants from State Center of Attention to Brain Injury were recruited.

Interventions: Patients were randomly assigned to 2 groups where the experimental group received sEMG-BFB for the upper trapezius and middle deltoid muscles of the upper limb with hemiparesis and the control group received a placebo of the same technique. Both treatments were applied for 6 weeks. The score of the Fugl-Meyer Assessment-Upper Extremity" for functionality and shoulder range of motion were objectified. Root mean square (RMS) value was assessed as a secondary measure Data were collected before and after intervention.

A protocol of sEMG-BFB in upper limb may have an important role in the recovery of subjects with upper limb hemiparesis.

ELIGIBILITY:
Inclusion Criteria:

* acquired brain injury after two months of medical evolution at least;
* suffer paretic upper limb;
* spasticity no greater than 3 in the modified Ashworth scale;
* minimum active ROM of 20º of glenohumeral abduction.

Exclusion Criteria:

* peripheral nerve injury, fractures of upper limb, cervical radiculopathy, complete luxation of the shoulder and severe cognitive impairment.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper-Extremity Scale (FMA-UE) | 15 minutes
  Assess functionality found in the motor recruitment of the paretic shoulder muscles after brain injury

SECONDARY OUTCOMES:
range of motion | 10 minutes
  Articular goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Maria Torres Lacomba, PhD, Study Director — University of Alcalá

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogan-Aslan M, Nakipoglu-Yuzer GF, Dogan A, Karabay I, Ozgirgin N. The effect of electromyographic biofeedback treatment in improving upper extremity functioning of patients with hemiplegic stroke. J Stroke Cerebrovasc Dis. 2012 Apr;21(3):187-92. doi: 10.1016/j.jstrokecerebrovasdis.2010.06.006. Epub 2010 Sep 29. PMID 20880720
- [Background] Giggins OM, Persson UM, Caulfield B. Biofeedback in rehabilitation. J Neuroeng Rehabil. 2013 Jun 18;10:60. doi: 10.1186/1743-0003-10-60. PMID 23777436
- [Result] De Baets L, Jaspers E, Janssens L, Van Deun S. Characteristics of neuromuscular control of the scapula after stroke: a first exploration. Front Hum Neurosci. 2014 Nov 17;8:933. doi: 10.3389/fnhum.2014.00933. eCollection 2014. PMID 25477805
- [Derived] Lirio-Romero C, Torres-Lacomba M, Gomez-Blanco A, Acero-Cortes A, Retana-Garrido A, de la Villa-Polo P, Sanchez-Sanchez B. Electromyographic biofeedback improves upper extremity function: a randomized, single-blinded, controlled trial. Physiotherapy. 2021 Mar;110:54-62. doi: 10.1016/j.physio.2020.02.002. Epub 2020 Feb 15. PMID 32718746